CLINICAL TRIAL: NCT06516835
Title: The Influence of Diluted and Undiluted Enteral Nutrition on Nutritional Tolerance in Critically Ill Patients After Gastrointestinal Surgery - a Randomized Controlled Trial
Brief Title: Diluted and Undiluted Enteral Nutrition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Collaborators: Nutricia Fundation (Unknown); Catholic University of Lublin (Unknown)
Responsible Party: Principal Investigator, Michał Borys, associate professor, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KE-0254/92/05/2024
Record Dates: First submitted 2024-07-07; First posted 2024-07-24 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Critical Illness; Surgery; Enteral Feeding Intolerance; Gastro-Intestinal Disorder; Quality of Life
Keywords: Zonulin; Intestinal fatty-acid binding protein (I-FABP); Ketones; Microbiome
MeSH Terms: conditions — Critical Illness; Digestive System Diseases; Ketosis

STUDY DESIGN:
Intervention Model Description: Two groups will be randomly allocated to ENF or IVF group
Who Masked: Participant
Masking Description: The patient will not be aware of the allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enteral nutrition fluid - ENF (Experimental): Enteral nutrition will be given continuously with glucose-Na-K Baxter 50 mg/ml solution for infusion (GNAK)-both products to the gastrointestinal tract in the same volume.
  Interventions: Other: Enteral fluid
- Intravenous fluid - IVF (Experimental): Enteral nutrition will be given continuously to the gastrointestinal tract. GNAK will be given continuously intravenously in the same volume.
  Interventions: Other: Intravenous fluid

INTERVENTIONS:
Other: Enteral fluid — GNAK will be administered to the gastrointestinal tract with EN in the same volume.
  Other Names: ENF
  Arms: Enteral nutrition fluid - ENF
Other: Intravenous fluid — Undiluted EN will be given to the gastrointestinal tract. GNAK, in the same volume, will be administered intravenously.
  Other Names: IVF
  Arms: Intravenous fluid - IVF

SUMMARY:
Adult patients after elective major abdominal surgeries who are planned to be admitted to the Intensive Care Unit (ICU) can be included in the trial.

Each patient will be fed via the gastrointestinal tract. Half of the patients will receive enteral nutrition (EN) with additional fluids, and the rest will receive undiluted EN.

The primary aim of this study is feeding intolerance assessment in both groups of patients.

DETAILED DESCRIPTION:
Approximately 50 % of the intensive care unit (ICU) population has feeding intolerance (FI), which includes nausea, vomiting, diarrhea, and others. Some studies suggest that FI can be alleviated in patients fed with supplemental parenteral nutrition (PN).

Adult patients after elective major abdominal surgeries who are planned to be admitted to the ICU can be included in the trial.

After the ICU admission, the patient will be stabilized, including warming, correction of water, electrolyte, and acid-base disorders, and blood transfusion if required. The fluid therapy will be monitored using the transpulmonary dilution technique.

Then, an attending physician will contact an investigator. The investigator will decide about the randomization (no contraindication). The investigators plan to maintain fluid therapy with continuous Glucose-Na-K Baxter 50 mg/ml solution for infusion (GNAK). GNAK will be administered in the same flow as EN, enterally or intravenously (i.v.).

Patients will be randomized to one of two studied groups:

* Continuous EN will be administered solely to the GI tract in the first group. The same dose of GNAK will be given i.v. (IVF group).
* In the second group, GNAK will be administered enterally with EN, a routine practice in our department (ENF group).

The attending physician will correct all fluid disturbances with balanced fluids or blood products according to laboratory tests and hemodynamic monitoring. GNAK will only be given as maintenance fluid with EN.

The primary outcome of our study will be feeding intolerance (FI).

FI is a composite outcome consisting of at least one of the following:

* Incidents of nausea and vomiting (nausea measured with a 4-point verbal descriptive scale (0=no nausea, 1=mild, 2=moderate, 3=severe))
* Incidents of diarrhea (≥ three loose stools per day)
* Increased gastric residual volume (> 500 ml of gastric aspirate/ 6 hours). Only in patients after lower GI tract surgeries (with intact stomach and gastric feeding)
* Achieving target EN on day three and later: 80% of protein requirements according to ESPEN (1.3/kg of ideal body weight (patients BMI < 30) or adjusted body weight, BMI ≥ 30)
* Administration of prokinetic agents. Starting with both erythromycin (125mg twice daily enterally) and metoclopramide (10mg three times per day i.v.)

Secondary outcomes (routinely performed procedures):

* PN requirements (days of support, grams of proteins, extra protein calories per day, contribution of PN in total nutrition)
* Insulin consumption (units per day and total per stay)
* Electrolyte supplementation (potassium, phosphorus, calcium, and magnesium in mmol/ stay)
* Enteral access obstruction (rinsing with fluid, need for replacement) per stay
* Intraabdominal pressure (twice daily)
* Sequential Organ Failure Assessment Score (twice daily)
* Fluid balance: additional fluids given intravenously during ICU stay
* Blood product transfusion
* Acute kidney injury, according to KDIGO definition
* Usage of vasoactive drugs: cumulative dose per stay
* Hemodynamic parameters, measured at least twice per day, such as stroke volume variation, pulse pressure variation, cardiac output, global end-diastolic volume, systemic vascular resistance, and extravascular lung water
* Laboratory tests, including lactate, electrolytes, arterial blood gas analysis, coagulation, total blood count
* Infections during the stay (site, antibiotics requirements)
* Mechanical ventilation time (hours)
* ICU stay (days)
* Hospital stay (days)
* Hospital mortality
* Intestinal fatty-acid binding protein (I-FABP) collection from blood and urine once daily during ICU stay
* Serum zonulin on the 1st day, 4th day, and at ICU discharge
* Serum ketones collection at ICU admission, 4th day, and discharge
* Gut microbiome collection at ICU admission and discharge

Follow-up:

• Quality of recovery - phone interview 30 days after randomization

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for major abdominal surgery requiring ICU admission
* Having access to the GI tract (gastric or jejunal)
* Planned to be fed enterally

Exclusion Criteria:

* Patients unable to give informed consent
* After emergency surgeries
* Without access to the GI tract
* Individuals with contraindications to EN, such as short bowel syndrome, uncompensated shock, acidosis (pH < 7.1; lactate > 5 mmol/l), bleeding from the upper GI tract, obstruction, intestinal ischemia, abdominal compartment syndrome
* Patients with symptomatic gastro-esophageal reflux
* Expected ICU stay < 3 days
* Pregnancy and lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants having nausea and vomiting | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Incidents of nausea and vomiting (nausea measured with a 4-point verbal descriptive scale (0=no nausea, 1=mild, 2=moderate, 3=severe))
Number of participants having diarrhea | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Incidents of diarrhea (≥ three loose stools per day)
Number of participants having increased gastric residual volume | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Increased gastric residual volume (> 500 ml of gastric aspirate/ 6 hours). Only in patients after lower GI tract surgeries (with intact stomach and gastric feeding)
Number of participants in whom target EN will not be achieved | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Achieving target EN on day three and later: 80% of protein requirements according to ESPEN (1.3/kg of ideal body weight (patients BMI < 30) or adjusted body weight, BMI ≥ 30)
Number of participants in whom prokinetic agents will be used | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Administration of prokinetic agents according to the intensivist discretion. Starting with both erythromycin (125 mg twice daily enterally) and metoclopramide (10mg three times per day i.v.)

SECONDARY OUTCOMES:
Days of support with PN | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Days of support with parenteral nutrition during the ICU stay.
Contribution of PN in total nutrition | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Percentage contribution of parenteral nutrition in total patient feeding understand as protein demands
Insulin consumption | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Insulin consumption - units per day and total per stay
Electrolyte supplementation | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Electrolyte supplementation - potassium, phosphorus, calcium, and magnesium in mmol/ stay
Enteral access obstruction | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Need for replacement outside the ICU or under endoscopy assistance. Number of such procedures per stay.
Intraabdominal pressure | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Intraabdominal pressure via urinary catheter twice daily
Sequential Organ Failure Assessment Score (SOFA) | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Calculating SOFA twice daily - from 0 to 24 - 0 means the lack of organ failure; 24 multiorgan failure
Fluid balance | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Additional crystalloids or colloids given intravenously during ICU stay measured in milliliters
Blood products transfusion | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Transfusion of any blood products, including red-packed cells, fresh-frozen plasma, platelets, and cryoprecipitate, measured in units per stay.
Acute kidney injury (AKI) | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Recognition of AKI according to Kidney Disease: Improving Global Outcomes (KDIGO) definition
Vasoactive drugs | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Usage of vasoactive drugs including noradrenaline, dobutamine, dopamine, adrenaline, and others measured in milligrams as cumulative dose per stay
Stroke volume variation | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Measurement of stroke volume variation presented in percent twice daily during the patient stay
Cardiac output | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Measurement of cardiac output (L/min) with pulmonary thermodilution technique twice daily during the patient's stay
Systemic vascular resistance | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Measurement of systemic vascular resistance (dynes/sec/cm-5) with pulmonary thermodilution technique twice daily during the patient's stay
Extravascular lung water | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Measurement of extravascular lung water index (ml/kg) with pulmonary thermodilution technique twice daily during the patient's stay
Lactates | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  At least once daily, arterial blood lactates (mmol/L) will be measured
Complete blood count (CBC) | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Once daily CBC will be tested
Blood proteins | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Plasma protein concentrations (g/dL) will measured at least once a week.
Infection site | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Site of infection during the ICU stay.
Antibiotics | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Antibiotics wchich will be used in ICU.
Blood albumins | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Plasma albumin concentrations (g/dL) will measured at least once a week.
C-reactive protein (CRP) | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  CRP (mg/L) will be measured once daily.
Procalcitonin (PCT) | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  PCT (ng/mL) will be measured once daily.
Mechanical ventilation | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Mechanical ventilation time in hours per stay
Intensive care unit (ICU) stay | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  ICU stay in days
Hospital stay | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Hospital stay in days
Hospital mortality | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  In-hospital mortality
Intestinal fatty-acid binding protein (I-FABP) | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  I-FABP concentrations (nmol/mL) will be measured in the blood and urine once daily.
Zonulin | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Zonulin concetration (ng/mL) will measured in the patient's blood on the 1st day, 4th day, and at the ICU discharge.
Ketones | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Serum ketone concentrations (mmol/L) will be collected and measured at ICU admission, 4th day, and discharge
Microbiome | From the date of randomization until the date of the ICU discharge or death but no longer than 8 weeks, whichever came first
  Intestinal microbiome collection upon admission and discharge from the ICU. Sequencing of the V3 V4 region of the 16SrRNA gene using NGS using Illumina technology, 2x250 bp, min. 100,000 readings, including DNA isolation. Preparation of the OTU table and basic alpha biodiversity measures
Quality of recovery | 30 days after randomization
  Phone interview using a modified version of Quality of recovery-40 scale (37-185 points,more points better) 30 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Michal Borys, MD, PhD, Principal Investigator — Medical University of Lublin
Locations (5):
- Poland (5):
  - Provincial Hospital in Gorzow Wielkopolski, Gorzów Wielkopolski
  - Fifth Military Hospital, Krakow
  - First Military Hospital, Lublin
  - II Department of Anesthesia and Intensive Care, Medical University of Lublin, Lublin
  - Provincial Hospital in Opole, Opole

IPD SHARING:
Plan to Share IPD: No